CLINICAL TRIAL: NCT05658276
Title: Establishing Physiologic Outcomes for Ventricular Unloading on VA ECMO
Status: Withdrawn | Type: Observational
Why Stopped: Did not enroll, prioritizing randomized trial.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Joseph Tonna, Associate Professor, Division of Cardiothoracic Surgery, University of Utah
Other Study IDs: 142543
Record Dates: First submitted 2022-10-31; First posted 2022-12-20 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-03

CONDITIONS: Cardiogenic Shock
Keywords: Mechanical circulatory support
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With LV Unloading: Adults (18+) who are in cardiogenic shock and being treated with mechanical circulatory support (veno-arterial ECMO) inserted peripherally. The patients in this group will also have an additional device, such as an Impella or an intra-aortic balloon pump (IABP) for left ventricular unloading. The decision whether or not to unload the patient will be purely clinical.
  Data will be collected from the patient's chart and entered into a secure database. A standard complete transthoracic echocardiogram will be completed at enrollment and then again 7 days from enrollment (+/- 2 days). Additional blood tests will be ordered for the 7 days after enrollment. All tests will be ordered on Day 1 (patient on ECMO, prior to any LV unloading) and additionally as follows:
  * Troponin: Daily for 7 days
  * NT-proBNP: Daily for 7 days
  * PCO2 gap (in blood gas analysis): Every 6 hours for 3 days
  * Lactate (in blood gas analysis): Every 12 hours for 3 days
  * cBIN1: Twice in 7 days
- Without LV Unloading: Adults (18+) who are in cardiogenic shock and being treated with mechanical circulatory support (veno-arterial ECMO) inserted peripherally. The patients in this group will not have any LV unloading device in addition to the ECMO support. The decision not to do LV unloading will be purely clinical.
  Data will be collected from the patient's chart and entered into a secure database. A standard complete transthoracic echocardiogram will be completed at enrollment and then again 7 days from enrollment (+/- 2 days). Additional blood tests will be ordered for the 7 days after enrollment. All tests will be ordered on Day 1 (patient on ECMO, prior to any LV unloading) and additionally as follows:
  * Troponin: Daily for 7 days
  * NT-proBNP: Daily for 7 days
  * PCO2 gap (in blood gas analysis): Every 6 hours for 3 days
  * Lactate (in blood gas analysis): Every 12 hours for 3 days
  * cBIN1: Twice in 7 days

SUMMARY:
Aim 1: Prospective, observational analysis of the association between echocardiographic measures of cardiac function and left ventricular unloading on VA ECMO.

Aim 2: Prospective, observational analysis of the association between clinical laboratory biomarkers and left ventricular unloading on VA ECMO.

DETAILED DESCRIPTION:
Mechanical circulatory support (MCS) is increasingly utilized as a means of hemodynamic support among cardiogenic shock (CS) patients refractory to optimal medical management. MCS modalities include using either an intra-aortic balloon pump (IABP), Impella®, or ECMO, each with unique benefit/harm profiles. Among the various MCS devices, extracorporeal membrane oxygenation (ECMO) is described as the highest level of support, capable of providing 5+ liters per minute of oxygenated blood flow but is the most invasive. Despite the benefit of maximal cardiopulmonary support, ECMO increases afterload in a failing heart. Left ventricular (LV) unloading or decompression (using simultaneous IABP or Impella®) has been suggested as potential improvement. Observational studies suggest a benefit with LV unloading during VA ECMO for CS, but the mechanisms underlying the association are poorly understood. Prior to trials, a mechanistic understanding of the effect of different LV unloading strategies on key physiologic abnormalities in CS is needed, as the physiologic effects of LV unloading during VA ECMO for CS remain insufficiently defined.

The objective of this study is to define serial changes in common clinical variables routinely obtained during management of patients in CS. These clinical variables are readily accessible to clinicians, but are not typically collected in a sufficiently granular serial manner to characterize their utility as clinical biomarkers. By obtaining scheduled assessments, repeated in a prospective cohort over the clinical course of CS, the investigators will define the physiologic effects of different LV unloading strategies in cardiogenic shock. We will examine a) echocardiographic measures of ventricular distension, and b) blood biochemical measures of peripheral perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years of age or older
* Patients with cardiogenic shock
* Patients with mechanical circulatory support, specifically veno-arterial extracorporeal membrane oxygenation (VA ECMO) inserted peripherally

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to our facility in cardiogenic shock.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Left ventricular function (ejection fraction) | Day 1/Enrollment
  Ejection fraction will be measured via echocardiogram and compared between time points and between groups
Left ventricular function (ejection fraction) | After LV unloading (within the first week of ECMO treatment; no specific day as this is a clinical decision)
  Ejection fraction will be measured via echocardiogram and compared between time points and between groups
Left ventricular function (ejection fraction) | Day 5
  Ejection fraction will be measured via echocardiogram and compared between time points and between groups

SECONDARY OUTCOMES:
Distension | Day 1/Enrollment
  Left ventricular end-diastolic dysfunction (LVEDD) will be measured via echocardiogram and compared between groups and between time points.
Distension | After LV unloading (within the first week of ECMO treatment; no specific day as this is a clinical decision)
  Left ventricular end-diastolic dysfunction (LVEDD) will be measured via echocardiogram and compared between groups and between time points.
Distension | Day 5
  Left ventricular end-diastolic dysfunction (LVEDD) will be measured via echocardiogram and compared between groups and between time points.
Peripheral perfusion per lactate | Daily (days 1-7)
  Measurements of lactate will indicate differences in peripheral perfusion between time points and between groups
Peripheral perfusion per CO2 gap | Daily (days 1-7)
  Measurements of carbon dioxide (CO2) gap will indicate differences in peripheral perfusion between time points and between groups
Cardiac injury per troponin | Daily (days 1-7)
  Measurements of troponin will indicate levels of cardiac injury between time points and between groups.
Cardiac injury per BNP | Daily (days 1-7)
  Measurements of B-type natriuretic peptide (BNP) will indicate levels of cardiac injury between time points and between groups.
Cardiac injury per cBIN1 | Twice in 7 days
  Measurements of cardiac BIN1 (cBIN1) will indicate levels of cardiac injury between time points and between groups.

CONTACTS AND LOCATIONS:
Locations (2):
- University of Utah, Salt Lake City, Utah, United States
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this time.

REFERENCES:
- [Background] Tonna JE, Selzman CH, Bartos JA, Presson AP, Ou Z, Jo Y, Becker L, Youngquist ST, Thiagarajan RR, Johnson MA, Rycus P, Keenan HT. The Association of Modifiable Postresuscitation Management and Annual Case Volume With Survival After Extracorporeal Cardiopulmonary Resuscitation. Crit Care Explor. 2022 Jul 25;4(7):e0733. doi: 10.1097/CCE.0000000000000733. eCollection 2022 Jul. PMID 35923595
- [Background] Rao P, Khalpey Z, Smith R, Burkhoff D, Kociol RD. Venoarterial Extracorporeal Membrane Oxygenation for Cardiogenic Shock and Cardiac Arrest. Circ Heart Fail. 2018 Sep;11(9):e004905. doi: 10.1161/CIRCHEARTFAILURE.118.004905. PMID 30354364
- [Background] Hitzeman TC, Xie Y, Zadikany RH, Nikolova AP, Baum R, Caldaruse AM, Agvanian S, Melmed GY, McGovern DPB, Geft DR, Chang DH, Moriguchi JD, Hage A, Azarbal B, Czer LS, Kittleson MM, Patel JK, Wu AHB, Kobashigawa JA, Hamilton M, Hong T, Shaw RM. cBIN1 Score (CS) Identifies Ambulatory HFrEF Patients and Predicts Cardiovascular Events. Front Physiol. 2020 May 25;11:503. doi: 10.3389/fphys.2020.00503. eCollection 2020. PMID 32670075
- [Background] Nikolova AP, Hitzeman TC, Baum R, Caldaruse AM, Agvanian S, Xie Y, Geft DR, Chang DH, Moriguchi JD, Hage A, Azarbal B, Czer LS, Kittleson MM, Patel JK, Wu AHB, Kobashigawa JA, Hamilton M, Hong T, Shaw RM. Association of a Novel Diagnostic Biomarker, the Plasma Cardiac Bridging Integrator 1 Score, With Heart Failure With Preserved Ejection Fraction and Cardiovascular Hospitalization. JAMA Cardiol. 2018 Dec 1;3(12):1206-1210. doi: 10.1001/jamacardio.2018.3539. PMID 30383171
- [Background] Eckman PM, Katz JN, El Banayosy A, Bohula EA, Sun B, van Diepen S. Veno-Arterial Extracorporeal Membrane Oxygenation for Cardiogenic Shock: An Introduction for the Busy Clinician. Circulation. 2019 Dec 10;140(24):2019-2037. doi: 10.1161/CIRCULATIONAHA.119.034512. Epub 2019 Dec 9. PMID 31815538
- [Background] Combes A, Price S, Slutsky AS, Brodie D. Temporary circulatory support for cardiogenic shock. Lancet. 2020 Jul 18;396(10245):199-212. doi: 10.1016/S0140-6736(20)31047-3. PMID 32682486
- [Background] Kim D, Jang WJ, Park TK, Cho YH, Choi JO, Jeon ES, Yang JH. Echocardiographic Predictors of Successful Extracorporeal Membrane Oxygenation Weaning After Refractory Cardiogenic Shock. J Am Soc Echocardiogr. 2021 Apr;34(4):414-422.e4. doi: 10.1016/j.echo.2020.12.002. Epub 2020 Dec 13. PMID 33321165
- [Background] Aissaoui N, Luyt CE, Leprince P, Trouillet JL, Leger P, Pavie A, Diebold B, Chastre J, Combes A. Predictors of successful extracorporeal membrane oxygenation (ECMO) weaning after assistance for refractory cardiogenic shock. Intensive Care Med. 2011 Nov;37(11):1738-45. doi: 10.1007/s00134-011-2358-2. Epub 2011 Oct 1. PMID 21965097

DOCUMENTS (1):
  • Informed Consent Form (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT05658276/ICF_000.pdf